CLINICAL TRIAL: NCT05566496
Title: The Findings of Resting-state Functional Magnetic Resonance Imaging, Diffusion Spectrum Imaging, and Wideband Magnetic Resonance Imaging in Subtypes of Tics-related Disorders
Brief Title: The Findings of Magnetic Resonance Imaging in Subtypes of Tics-related Disorders
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201503062RIND
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Tourette Syndrome in Children
Keywords: MRI; pediatric neurology

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tourette: Age less than 18 years old Diagnosed as Tourette syndrome or chronic tic disorders No other neuropsychiatric disorders
  Interventions: Diagnostic Test: Brain MRI
- Healthy: Age less than 18 years old No other neuropsychiatric disorders
  Interventions: Diagnostic Test: Brain MRI

INTERVENTIONS:
Diagnostic Test: Brain MRI — All participants receive brain MRI evaluation and clinical evaluation of tic severity.

SUMMARY:
The findings of resting-state functional magnetic resonance imaging and diffusion spectrum imaging in subtypes of tics-related disorders

ELIGIBILITY:
Inclusion Criteria:

* Age less than 18 years old
* Diagnosed as Tourette syndrome or chronic tic disorders

Exclusion Criteria:

* History of neuropsychiatric disorders
* Already receive treatment for Tourette syndrome/chronic tics disorder
* Have some device not allowed for MRI scan

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: We enrolled treatment-naive Tourette syndrome or chronic tic disorder pediatric patients for Tourette group and healthy age- and gender-matched participants for healthy control
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-10-20 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Difference between healthy and Tourette group | 2 years after enrollment for primary evaluation
  Difference of MRI result between healthy and Tourette group

CONTACTS AND LOCATIONS:
Overall Officials: Wang-Tso Lee, Principal Investigator — National Taiwan University Children Hospital Pediatric neurology department
Locations (1):
- National Taiwan University Children Hospital Pediatric Neurology Department, Taipei, Taiwan